CLINICAL TRIAL: NCT01056432
Title: Phase I Study of Portable Bone Ultrasonometer for Osteoporosis Assessment
Brief Title: Bone UltraSonic Scanner (BUSS) Clinical Optimization Study
Acronym: BUSS
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: BUSS-02; 2R44AG017400 (NIH)
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis, bone fracture risk, bone ultrasonometry
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this clinical study using Bone UltraSonic Scanner (BUSS) is to obtain clinical data which will help to optimize the BUSS examination procedure and its diagnostic algorithms for assessment of bone conditions.

DETAILED DESCRIPTION:
The specific aims of this clinical study are:

1. To optimize the data collection technique and establish an examination procedure;
2. To collect data necessary for assessing the performance of BUSS sensors;
3. To evaluate the probe ergonomic design and participant tolerance to probe application;
4. To assess the clinical suitability of the software interface in data collection;
5. To adjust the BUSS diagnostic algorithms using dual-energy X-ray absorptiometry (DEXA) data as a "gold" standard in osteoporosis detection and characterization;
6. To evaluate BUSS performance including ease of use and consistency.

ELIGIBILITY:
Inclusion Criteria:

Any race or ethnical group DEXA examination scheduled within next two weeks or DEXA examination was completed within the last six months adn DEXA results are available

Exclusion Criteria:

Open wounds or rashes on the tibial testing area Active skin infection Recent tibia surgery Abnormal tibia Anatomy Current or previous tibial fracture Body Mass Index >34.9 Hyperparathyroidism or hypoparathyroidism within 5 years Osteitis deformans Renal osteodystrophy Osteomalacia Stroke with total or partial paralysis with residual disability lasting more than 3 months Current or recent (within past 6 months) use of bone-active drugs Drugs under research protocols Chronic use of over the counter antacids

-

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will consist of groups with no history of osteoporosis, established osteoporosis and may include documented history of fracture.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To obtain clinical data which will help to optimize the BUSS examination procedure and its diagnostic algorithms for assessment of bone conditions. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, Ph.D., D.Sc., Principal Investigator — Artann Laboratories
Locations (1):
- Health Smart Medical Center, Philadelphia, Pennsylvania, United States